CLINICAL TRIAL: NCT06117085
Title: First Clinical Feasibility Study Using the CellFX® Percutaneous Electrode (PE) System for the Treatment of Symptomatic Benign Thyroid Nodules
Brief Title: CellFX ® Percutaneous Electrode (PE) Treatment of Symptomatic Benign Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulse Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP-TF-024
Record Dates: First submitted 2023-10-26; First posted 2023-11-03 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Thyroid Nodule (Benign)
MeSH Terms: conditions — Thyroid Nodule | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Percutaneous Treatment Arm (Experimental): CellFX Percutaneous Treatment under ultrasound guidance using nanosecond Pulse Field Ablation (nsPFA)
  Interventions: Device: CellFX® Percutaneous Electrode (PE) System

INTERVENTIONS:
Device: CellFX® Percutaneous Electrode (PE) System — Percutaneous treatment with CellFX® Percutaneous Electrode using nanosecond pulse field ablation (nsPFA) technology

SUMMARY:
The objective of this clinical feasibility study is to evaluate initial clinical safety and device performance of the CellFX Percutaneous Electrode (PE) System for the treatment of symptomatic benign thyroid nodules.

DETAILED DESCRIPTION:
Cohort 1: (CellFX PE Procedure and Surgery) The first five enrolled subjects will be patients with planned thyroidectomy. The site investigator will perform the CellFX procedure followed by an ultrasound evaluation. The site investigator will then perform a partial or total thyroidectomy. Tissue samples from the CellFX targeted treated areas will be sent to the pathology lab for gross and histological evaluation. The participant will exit the study on the same day of surgery.

Cohort 2: (CellFX PE Procedure with 12 months follow-up) When Cohort 1 is completed, up to 25 subjects will undergo a CellFX treatment using a percutaneous approach under ultrasound guidance. After CellFX treatment, all subjects will be followed weekly until 1 month, 3 months, 6 months and 12 months post-CellFX PE procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 or no older than 80 years of age
* Participant gives voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
* Participant must comply with study procedures including all follow-up visits diagnosis of thyroid nodule confirmed by ultrasonography ≤Grade 3 (2017 ACR TI-RADS and fine needle aspiration biopsy FNA (Bethesda category II ) with no macro-calcifications in target nodule within 30 days of enrollment
* Participant has single nodule ≤ 6.0 cm in greatest dimension.
* Participant may have abnormal thyroid function, such as suppressed thyrotropin (TSH) levels, at the screening visit
* Participant has no abnormal cervical lymph nodes during screening visit examination
* Participant has thyroid nodule causing appearance, pressure or swallowing symptoms
* Participant has absence of abnormal vocal cord mobility by ultrasound evaluation

Exclusion Criteria:

* Participant has an implantable electronic medical device. (i.e., pacemaker, implantable cardioverter defibrillator)
* Participant has an active systemic infection on the day of the CellFX PE procedure with either fever, leukocytosis or requiring intravenous antibiotics or history of head and neck, pulmonary or systemic infection in the last 2 weeks prior to CellFX PE procedure
* Participant is known to be immune compromised
* Participant is a member of a vulnerable population including individuals employed by the Sponsor, clinic site, or entity associated with the conduct of the study
* Participant had previous neck irradiation
* Participant has history of familial thyroid cancer in more than two first-degree relatives
* Participants currently suffering from hematological diseases or bleeding tendency, or patients currently requiring continuous administration of antiplatelet and anticoagulant drugs
* Ultrasonographic evidence of calcifications, irregular margins or sonographic features that are suspicious for malignancy
* Nodule likely to be in contact with the recurrent laryngeal nerve on ultrasound evaluation
* History of cardiac arrhythmia, uncontrolled hypertension, liver or kidney disease, or recent history of myocardial infarctions or structural heart disease as determined by the Investigator
* History of a coagulation mechanism disorder or bleeding tendency
* Abnormal contralateral vocal cord function
* Allergy or contraindication to assigned analgesia/anesthesia
* Females of childbearing potential who are nursing, pregnant, or planning to become pregnant during the study period
* Have any condition or situation which, in the Investigator's opinion, puts the participant at significant risk, could confound the study results, or may interfere significantly with the participant's participation in the study
* Use of any other investigational drug, therapy, or device within 30 days prior to enrollment or concurrent participation in another research study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with serious adverse device effects | 1 month, 3 months, 6 months and 12 months post-CellFX PE procedure
  The primary safety endpoint will be assessed by the incidence of serious adverse device effects
Number of Participants with Acute nodular volume loss | 6 months post-CellFX PE procedure
  Acute procedural success defined as a ≥ 50% nodule volume loss by ultrasonography and without serious adverse device effects within 6-months of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Prof Stefano Spiezia, MD, Principal Investigator — Chief of Endocrine and Ultrasound Guided Surgery, Operative Unit
Locations (1):
- Ospedale del Mare | ASLNA1 Centro, Naples, Italy

IPD SHARING:
Plan to Share IPD: No